CLINICAL TRIAL: NCT06155591
Title: Effectiveness of the Community Nurse Case Manager in Primary Care for Complex and Pluripathological Chronic Dependent Patients: Study Protocol
Brief Title: Case Management of Complex Pluripathology in Primary Care
Acronym: ENGESCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: José Ignacio Recio Rodriguez (Other)
Collaborators: Consejo General de Colegios Oficiales de Enfermería de España (Unknown); Instituto Español de Investigación Enfermera (Unknown); Gerencia Regional de Salud de Castilla y Leon (Other)
Responsible Party: Sponsor-Investigator, José Ignacio Recio Rodriguez, Full Professor at the University. PhD, University of Salamanca
Organization: University of Salamanca (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GRS 2490/B/22
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Complex and Chronic Pluripathology
Keywords: Multimorbidity; Functional Dependence; Case Management; Primary Health Care; Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Usual care of complex and pluripathological chronic patients (CPCP)
- Experimental Group (Experimental): Usual care of CPCP + Community Nurse Case Manager (CNCM) standardized protocol
  Interventions: Other: Community Nurse Case Manager (CNCM)

INTERVENTIONS:
Other: Community Nurse Case Manager (CNCM) — Their action protocol has been designed and sequenced according to the circumstances in which the Complex and Pluripathological Chronic Patient finds themself:
  * Pre-hospital discharge. The hospital Nurse Case Manager (HNCM) will contact the CNCM to inform of the imminent hospital discharge.
  * Hospital discharge: A comprehensive nursing assessment of the CPCP based on Marjory Gordon's functional patterns will be carried out.
  * Planned visits: An infographic will be provided to identify signs and symptoms of decompensation/exacerbation and a direct dial telephone number.
  * Proactive telephone follow-up: The CNCM will make comfort calls every week for the first month, every 15 days until the 3-months visit and every month until the 6- and 12-months visits.
  * Exacerbations/decompensations: An appointment will be arranged with their Primary Care physician.
  * Hospital readmission: The CNCM will be kept informed of the process through the HNCM and CPCP's digital clinical history.
  Arms: Experimental Group

SUMMARY:
Aims

To assess the effect of the implementation of the Community Nurse Case Manager (CNCM) in the care of complex and pluripathological chronic patients (CPCP) with dependence, from Primary Care, on functional capacity, cognitive performance, quality of life, consumption of health resources, clinical parameters, overload of the main caregiver, and satisfaction of the user and/or caregiver.

Design

Pre- and post-intervention quasi-experimental study in CPCP.

Methods

212 subjects will be recruited from two urban health centers in Salamanca (Spain) with complex and chronic pluripathology (CCP) associated to cardiac, respiratory pathology and/or diabetes mellitus, who are dependent and have a planned hospital discharge.

An initial evaluation will be performed after hospital discharge in both groups, including: anamnesis (prescribed drugs and symptoms attributable to the underlying pathology), physical examination (blood pressure, heart rate and oxygen saturation), determination of capillary HbA1c, and assessment of functional capacity (Barthel), cognitive performance (MoCA), quality of life (COOP-WONCA), therapeutic adherence and overload of the main caregiver (Zarit). There will be another evaluation at 3,6 and 12 months, when these same variables will be collected, in addition to the number of readmissions in each period and the satisfaction of the user and/or caregiver (Satisfad 14). The nurse from the Primary Care team will provide both groups with the usual care contemplated for this type of patient in the Portfolio of Services of the Health Service of Castilla y León. Additionally, in the experimental group there will be telephone follow-up and the caregiver will be trained on the signs of decompensation and the care required.

Conclusion

The deployment of the NCM (Nurse Care Manager) in Primary Care will provide comprehensive and individualized care to the CPCP and the main caregiver with proactive monitoring. In addition, it will reinforce the involvement of the caregiver and the patient to improve their self-care and will detect early signs and symptoms of decompensation to avoid hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Dependent complex and pluripathological chronic patients (CPCP) with associated cardiac and/or respiratory pathologies and/or diabetes mellitus
* Frail ≥1 point
* Require a main caregiver to perform basic activities of daily living (ABVD)
* Barthel ≤60 points and/or grade II or III dependency recognised by Social Services
* Are immobilised at home and/or require social resource management
* Agree to sign (themselves or their legal guardians) the informed consent for participation in the study

Exclusion Criteria:

* Patients with other pathologies associated with complex pluripathology
* With non-habitual caregivers
* Barthel ≥60 points or grade I dependency recognised by Social Services
* Who reside outside the area assigned to the Garrido Sur and Miguel Armijo health centres despite being assigned to them

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Activities of daily living | 0,1,3,6,12 months
  Evaluated by Barthel index. Score (0-100). A person is considered totally dependent if it is ˂20 points; severely dependent if it is between 25-60 points; moderately dependent if it is between 65-90 points; and mildly dependent if it is equal to 95 points
Cognitive performance | 0,3,6,12 months
  Evaluated by Montreal Cognitive Assessment (MoCA). Score (0-30). A score of 26 or higher is considered normal
Health-related quality of life | 0,3,6,12 months
  Evaluated by Health-related quality of life (COOP-WONCA test). This consists of a drawing representing a level of functioning on seven areas with a 5-level Likert scale. Higher scores express worse levels of functioning/well-being.

SECONDARY OUTCOMES:
Frailty | 0,1,3,6,12 months
  Evaluated by FRAIL questionnaire. This consists of 5 simple questions on fatigue, endurance, ambulation, comorbidity and weight loss. Persons scoring 1 point or more are considered frail
Primary caregiver overload | 0,3,6,12 months
  Evaluated by the Zarit scale. Score (22 - 110). A score ≥47 points being considered overburden
Therapeutic adherence | 1,3,6,12 months
  Evaluated by a scale to assess the patient's skills and knowledge of the prescribed treatment, adapted from the DRUGS and Med-Take scales. A score > 75%, the patient is adherence to treatment.
User satisfaction | 1,3,6,12 months
  Evaluated by Satisfad Questionnaire 14. Score (0-42). Each item is assessed through a 4-level Likert scale. A higher score means a higher level of satisfaction
Degree of dyspnoea | 0,1,3,6,12 months
  Evaluated by modified Medical Research Council Scale. This consists of 5 levels. The higher the level, the lower the tolerance to activity due to dyspnoea
Symptoms attributable to heart disease | 0,1,3,6,12 months
  Evaluated by the New York Heart Association Functional Classification. This consists of 4 Class. Class I patients have no symptoms, while those in classes II, III and IV have mild, moderate and severe symptoms, respectively
Number of hospital admissions | 1,3,6,12 months
  Collected from the patient's medical history
Number of drugs chronically prescribed | 0,1,3,6,12 months
  Collected from the patient's medical history
Weight | 0 months
  Collected from the patient's medical history
Height | 0 months
  Collected from the patient's medical history
Body mass index | 0 months
  Collected from the patient's medical history
Blood pressure systolic and diastolic | 0,1,3,6,12 months
  Measured in mmHg
Oxygen saturation | 0,1,3,6,12 months
  Measured in %
Heart rate | 0,1,3,6,12 months
  Measured in bpm
Capillary blood glucose | 0,1,3,6,12 months
  Measured in mg/dl
Capillary glycosylated haemoglobin | 0,3,6,12 months
  Measured in %

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iglesias-Sierra V, Sanchez-Aguadero N, Recio-Rodriguez JI, Sanchez-Salgado B, Garcia-Ortiz L, Alonso-Dominguez R. Effectiveness of the Community Nurse Case Manager in Primary Care for Complex, Pluripathological, Chronic, Dependent Patients: A Study Protocol. Nurs Rep. 2025 May 29;15(6):191. doi: 10.3390/nursrep15060191. PMID 40559482